CLINICAL TRIAL: NCT02403362
Title: A Phase 2, Open-Label, Multi-Center , Dose-Ranging Study of the Safety and Efficacy of Pegol-Sihematide (EPO-018B) for the Treatment of Anemia in Patients With Chronic Kidney Disease Not Requiring Dialysis.
Brief Title: Safety & Efficacy of EPO-018B for the Treatment of Anemia in Participants With Chronic Kidney Diseases Not on Dialysis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HS-EPOP2b
Record Dates: First submitted 2015-02-12; First posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Renal Failure; Chronic Kidney Disease; Anemia
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- EPO-018B 0.025 mg/kg (Experimental): EPO-018B starting dose of 0.025 milligram per kilogram (mg/kg) administered subcutaneously (SC) once every 4 weeks (Q4W) for a total of 6 doses
  Interventions: Drug: EPO-018B
- EPO-018B 0.05 mg/kg (Experimental): EPO-018B starting dose of 0.05 milligram per kilogram (mg/kg) administered subcutaneously (SC) once every 4 weeks (Q4W) for a total of 6 doses
  Interventions: Drug: EPO-018B
- EPO-018B 0.08 mg/kg (Experimental): EPO-018B starting dose of 0.08 milligram per kilogram (mg/kg) administered subcutaneously (SC) once every 4 weeks (Q4W) for a total of 6 doses
  Interventions: Drug: EPO-018B

INTERVENTIONS:
Drug: EPO-018B

SUMMARY:
The purpose of this study is to evaluate the safety,efficacy， pharmacodynamics (PD), and pharmacokinetics (PK) of multiple intravenous doses of EPO-018B in participants with chronic kidney disease (CKD) Who are not on dialysis

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥18 and≤70.
2. Chronic renal diseases stage 3 or 4 (estimated Glomerular Filtration Rate (eGFR) between 15 and 60 ml/min per 1.73 m2 using the CKD-EPI equation) and no expected need for dialysis during the study.
3. Patients who have not received any erythropoietic agents within 6 weeks prior to the first study dose.
4. Two hemoglobin values of ≥ 6.0 and < 10.0 g/dL at Screening
5. Patients with a transferrin saturation ≥ 20% or a ferritin ≥ 100 ng/mL. vitamin B12 and folic acid level above lower limit of normal.
6. Signed informed consent.

Exclusion Criteria:

1. Pregnant or lactating females.
2. Red blood cell transfusion within 3 months prior to study drug administration.
3. Known intolerance to any erythropoiesis stimulating agent (ESA) or pegylated molecule or to all parenteral iron supplementation products .
4. Hemolytic syndromes or coagulation disorder.
5. Hematological disease (including but not limited to myelodysplastic syndrome, hematological malignancy, hemoglobinopathy, pure red cell aplasia).
6. Chronic, uncontrolled, or symptomatic inflammatory disease (e.g., rheumatoid arthritis, systemic lupus erythematosus, etc.).
7. C reactive Protein (CRP)level greater than 30 mg/L within the 4 weeks prior to study drug administration.
8. Uncontrolled or symptomatic secondary hyperparathyroidism(iPTH>500pg/ml).
9. Poorly controlled hypertension within 2 weeks prior to study drug administration, per investigator's clinical judgment (e.g. systolic ≥ 160mm Hg, diastolic ≥ 100 mm Hg)
10. Chronic congestive heart failure (New York Heart Association Class IV).
11. Significant symptom within 6 months prior to study drug administration (e.g. myocardial infarction, serious or precarious coronary artery disease,stroke, respiratory disease, autoimmune disease, neuropathy, phrenopathy, hepatopathy including Active hepatitis B, Active hepatitis C, or ALT> 3 x upper limit of normal (ULN), AST> 3 x upper limit of normal (ULN), etc.).
12. A positive test for HIV antibody.
13. Tumor malignancy.
14. Expected survival less than 12 months.
15. Major surgery (may Massive bleeding) during the study.
16. Expected conception within 4 Weeks after the end of the Study Treatment.
17. The subject has participated in other clinical trial within the 6 weeks prior to study drug administration.
18. Have any other condition or prior therapy that, in the investigator's opinion, would make the subject unsuitable for the study, or unable or unwilling to comply with the study procedures.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who achieved a target hemoglobin response during the study | Baseline to Week 24
  A target hemoglobin response is defined as a hemoglobin increase of ≥ 1.0 gram per deciliter (g/dL) from baseline and a hemoglobin value ≥ 10.0 g/dL during the study

SECONDARY OUTCOMES:
Percentage of participants who response to study drug | Baseline to Week 24
  Hemoglobin response is defined as a hemoglobin increase of ≥ 1.0 gram per deciliter (g/dL) from baseline during the study
Average reticulocytes change from baseline | Baseline to Week 24
Average hemoglobin change from baseline | Baseline to Week 24
Incidence of adverse events | Baseline to Week 24
Incidence of serious adverse events | Baseline to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Xueqing Yu, Study Chair — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China